CLINICAL TRIAL: NCT06748326
Title: Laparoscopic Reduction of Intussusception in Children: Role in Primary Reduction After Failed Non-Surgical Therapies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelrahman Ahmed Khalil, Resident doctor at surgical department at Assiut university, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopy in Intussusception
Record Dates: First submitted 2023-11-12; First posted 2024-12-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Intussusception
MeSH Terms: conditions — Intussusception | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Children with intussusception that failed non surgical procedures and whose with recurrence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic reduction of intussusception in children (Other): The abdomen is insufflated through an umbilical ring incision and a trocar is inserted to act as a camera Port. Two other ports for manipulation are placed depend on the position of the intussusception either in the right lower quadrant and the left upper quadrant or both the upper left and lower left quadrants of the abdomen. These ports position is assuming that radiological reduction has carried the intussusceptum to the right colon. Two atraumatic bowel clamps are used for bowel manipulation. The reduction is achieved by traction placed on the proximal bowel (intussusceptum) out of the distal segment (the intussuscepien).
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Intussusception reduction by laparoscopy in children in failed non surgical procedures and in recurrence

SUMMARY:
Laparoscopic Reduction of Intussusception in Children: Role in Primary Reduction after Failed Non-Surgical Therapies.

DETAILED DESCRIPTION:
Intussusception is one of the main abdominal emergencies in children. Its diagnosis is usually based on the clinical features and confirmed either by U/S and /or barium enema and CT scan in rare occasion. Since the introduction of the hydrostatic reduction of intussusceptions by Ravitch in 1848, it became the gold standard management. However surgical intervention is required if this and other non-operative approaches fail. This typically involves 10 to 20% of cases. Early on, the approach has been through an open laparotomy and manual reduction of intussusception. Later, the introduction of the laparoscopy in the paediatric surgical field has added another dimension to the management of intussusception. In addition to its confirmed general benefits of less pain, better cosmoses, and low long-term risk of adhesive bowel obstruction, it also can be a diagnostic modality in certain cases, primary reduce the intussusception and in some cases to resect the pathological lead point or the damaged segment of bowel. The laparoscope allowed the surgeons to avoid unnecessary open procedures in cases of spontaneous reduction following enema reductions, obviating the need for an open procedure in up to 30% of cases. Despite of all mentioned above, its effectiveness has been questioned.

ELIGIBILITY:
Inclusion Criteria:

* 1. childs aged 1 year to 12 years with intussusception who failed the hydrostatic reduction.

Exclusion Criteria:

- 1. Childs with Bad general conditions ( coagulopathy, haemodynamic instability, and severe cardiopulmonary diseases).

2. Known primary disease e.g. lymphoma and major congenital anomalies. 3. Previous abdominal surgeries.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-05-03 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Results of Laparoscopy using in reduction of intussusception in children. | 6 months
  According to hospital stay, cosmesis and as a minimally invasive approach.